CLINICAL TRIAL: NCT06849089
Title: Holmium Laser Enucleation of the Prostate: Learning Curve Analysis and Comparison With TURP
Brief Title: HoLEP: Learning Curve Analysis and Comparison With TURP
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tarik Emre Sener, Associate Professor of Urology., Marmara University
Other Study IDs: MAR.UAD.0020
Record Dates: First submitted 2025-02-19; First posted 2025-02-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Prostatic Hyperplasia, Benign; Prostatic Obstruction
Keywords: prostate; prostatectomy; laser
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 - TURP patients: The last 100 patients who underwent bipolar TURP by the same surgeon who performed the HoLEP procedures in the study.
  Interventions: Procedure: Transurethral resection of prostate (TURP)
- Group 2 - Initial HoLEP patients: The initial 50 patients who underwent HoLEP, who were considered to be operated in the learning curve of the surgeon.
  Interventions: Procedure: Holmium laser enucleation of prostate
- Group 3 - Subsequent HoLEP patients: The subsequent 50 patients who underwent HoLEP, who were considered to be operated in the expert phase of the surgeon.
  Interventions: Procedure: Holmium laser enucleation of prostate

INTERVENTIONS:
Procedure: Transurethral resection of prostate (TURP) — The surgical intervention used to resect the benign adenomatous hyperplastic nodules of the prostate that cause obstruction and consequently lower urinary tract symptoms. The procedure uses a hot loop shaped knife, operated by electrocautery, to cut the obstructing tissues from center towards periphery of the prostate until the prostatic capsule is reached.
  Groups: Group 1 - TURP patients
Procedure: Holmium laser enucleation of prostate — The surgical intervention used to enucleate the benign adenomatous hyperplastic nodules of the prostate that cause obstruction and consequently lower urinary tract symptoms. The procedure uses a laser fiber to dissect the obstructing adenoma from the prostatic capsule starting from the plane in-between the capsule and the adenoma, meaning removal of tissues from periphery towards the center of the prostate.
  Groups: Group 2 - Initial HoLEP patients; Group 3 - Subsequent HoLEP patients

SUMMARY:
This study evaluates the outcomes of Holmium laser enucleation of the prostate (HoLEP) during both the learning and expert phases compared to transurethral resection of the prostate (TURP) in managing benign prostatic obstruction (BPO)-related lower urinary tract symptoms (LUTS). A prospective analysis of 200 men was conducted, dividing them into three groups: TURP (n=100), HoLEP during the learning curve (n=50), and HoLEP post-learning curve (n=50). Key outcomes assessed included the learning curve, perioperative safety, efficacy, functional recovery (IPSS, QoL, Qmax, PVR), surgical efficiency, and complication rates.

DETAILED DESCRIPTION:
INTRODUCTION Benign prostatic obstruction (BPO) is a common urological issue that leads to lower urinary tract symptoms (LUTS). BPO is typically caused by benign prostatic hyperplasia (BPH), a histopathological condition that contributes to BPO through two mechanisms: a static component, where the enlarged prostate tissue obstructs urine flow, and a dynamic component, where increased smooth muscle tone increases resistance to urinary flow. These changes can lead to LUTS, recurrent urinary tract infections, urinary retention, and hematuria.

LUTS due to BPO can be managed through conservative measures, pharmacological treatments, or surgical interventions. While conservative and pharmacological therapies offer temporary, symptom-based relief, surgical treatments aim to provide a more permanent solution. Transurethral resection of the prostate (TURP) has been the gold standard surgical treatment for BPO for many years. However, advances in laser technology and surgical techniques have led to the increased popularity of anatomical endoscopic enucleation of the prostate (AEEP) using lasers such as holmium yttrium-aluminum-garnet (YAG), thulium YAG, or thulium fiber laser in the past decade. HoLEP is quite versatile in achieving complete anatomic enucleation of prostate adenoma which provides a permanent relief of obstruction and prevents re-growth of remnant prostatic tissue.

The scientific evidence supports the superiority of HoLEP compared to TURP, which has long been the gold standard. However, HoLEP is not an easy surgical method to learn and expertise. The learning curve is a critical consideration in HoLEP, which requires significant technical skill and experience to achieve proficiency and optimal outcomes. Perioperative and postoperative variables are evaluated to assess surgeon performance over consecutive cases.

The learning curve has been reported to be variable in different studies showing results between 25 to 80 cases in different cohorts.

In this study, we aimed to evaluate the outcomes of HoLEP during both the learning curve and expert periods, and to compare these results with the long-established gold standard, TURP.

METHODS Eligible patients were men >50 years of age presenting to our outpatient clinic with LUTS attributed to BPO with an indication for surgical treatment according to EAU Guidelines on Non-Neurogenic Male Lower Urinary Tract Symptoms 14 and who underwent either TURP or HoLEP. Patients with a prior history of BPE surgery, history of prostate cancer diagnosis were excluded.

Patients who underwent HoLEP by a single surgeon were included in the study. HoLEP patients were divided into 2 groups. The initial 50 patients who underwent HoLEP were considered to be operated in the learning curve of the surgeon. The subsequent 50 patients who underwent HoLEP by the same surgeon were considered to be operated in the expert phase of the surgeon. For comparison with the TURP outcomes, the last 100 patients who underwent bipolar TURP by the same surgeon were included in the study.

TURP patients were grouped as Group 1, initial 50 HoLEP patients were grouped as Group 2 and the subsequent 50 HoLEP patients were grouped as Group 3.

Patients who had a urinary tract infection prior to surgery were treated with appropriate antibiotics according to the preoperative urine culture. All the patients were scheduled for surgery when a sterile urine culture was obtained. All the patients received second generation cephalosporins as prophylactic antibiotics prior to surgery according to the local institution's Infections Committee protocol. Bridging with low molecular weight heparin was performed for all the patients who were under anticoagulant or antiaggregant therapies.

The primary objective was to evaluate the success rate. The evaluated parameters were scores on International Prostate Symptom Score (IPSS) and Quality of Life (QoL) questionnaire, maximum urinary flow rate (Qmax) on uroflowmetry and post-void residual urine volume (PVR) and operation duration, surgical efficiency and learning curve of HoLEP using the Cumulative Sum (CUSUM) analysis, for which, enucleation efficiency was used as evaluated parameters.

The secondary objective was to evaluate the safety profile by comparing the postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* men >50 years of age
* presenting to our outpatient clinic with lower urinary tract symptoms attributed to benign prostatic obstruction
* indication for surgical treatment according to EAU Guidelines on Non-Neurogenic Male Lower Urinary Tract Symptoms

Exclusion Criteria:

* prior history of BPE surgery
* history of prostate cancer diagnosis

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men >50 years of age with with lower urinary tract symptoms due to benign prostatic obstruction
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Surgical efficiency | Perioperative/Periprocedural
  Surgical efficiency is defined as the resected / enucleated tissue volume in grams divided by total operation duration in minutes. The unit is g/min.
Preoperative International Prostate Symptom Score (IPSS) | Baseline
  The International Prostate Symptom Score (IPSS) is a standardized questionnaire used to assess the severity of lower urinary tract symptoms (LUTS) associated with benign prostatic obstruction (BPO). It consists of seven questions evaluating urinary symptoms (incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia) and one additional question on quality of life (QoL). Each symptom is rated on a scale from 0 to 5, with a total score ranging from 0 to 35, where higher scores indicate more severe symptoms.
Postoperative International Prostate Symptom Score (IPSS) | 6 months
  The International Prostate Symptom Score (IPSS) is a standardized questionnaire used to assess the severity of lower urinary tract symptoms (LUTS) associated with benign prostatic obstruction (BPO). It consists of seven questions evaluating urinary symptoms (incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia) and one additional question on quality of life (QoL). Each symptom is rated on a scale from 0 to 5, with a total score ranging from 0 to 35, where higher scores indicate more severe symptoms.
Preoperative Quality of Life (QoL) | Baseline
  The Quality of Life (QoL) question at the end of the International Prostate Symptom Score (IPSS) assesses how bothersome a patient's urinary symptoms are in daily life. It asks:
  Patients rate their response on a scale from 0 to 6, where 0 = delighted and 6 = terrible, providing a subjective measure of symptom impact on overall well-being.
Postoperative Quality of Life (QoL) | 6 months
  The Quality of Life (QoL) question at the end of the International Prostate Symptom Score (IPSS) assesses how bothersome a patient's urinary symptoms are in daily life. It asks:
  Patients rate their response on a scale from 0 to 6, where 0 = delighted and 6 = terrible, providing a subjective measure of symptom impact on overall well-being.
Preoperative Maximum urinary flow rate (Qmax) on uroflowmetry | Baseline
  Maximum urinary flow rate (Qmax) is the highest flow rate of urine (measured in milliliters per second, mL/s) recorded during uroflowmetry, a non-invasive test that assesses urinary flow dynamics.
PostoperativeMaximum urinary flow rate (Qmax) on uroflowmetry | 6 months
  Maximum urinary flow rate (Qmax) is the highest flow rate of urine (measured in milliliters per second, mL/s) recorded during uroflowmetry, a non-invasive test that assesses urinary flow dynamics.
Operation duration | Perioperative/Periprocedural
  Operation duration refers to the total time taken to complete a surgical procedure, typically measured from the instrument insertion to the completion of the surgery. In the context of HoLEP and TURP, it includes steps such as enucleation (for HoLEP), resection (for TURP), hemostasis, and tissue morcellation (for HoLEP)
Learning curve | through study completion, an average of 6 months
  The learning curve represents the time and number of cases required for a surgeon to achieve proficiency in a procedure, balancing efficiency, safety, and outcomes.

SECONDARY OUTCOMES:
Complication rate | through study completion, an average of 6 months
  Complication rate refers to the frequency of adverse events occurring during or after a surgical procedure, typically expressed as a percentage of total cases.
Incontinence rate | through study completion, an average of 6 months
  Incontinence rate refers to the proportion of patients experiencing urinary incontinence after surgery, typically expressed as a percentage of total cases.
Urethral stricture rate | through study completion, an average of 6 months
  Urethral stricture rate refers to the proportion of patients who develop a narrowing of the urethra following a surgical procedure, expressed as a percentage of total cases.

CONTACTS AND LOCATIONS:
Overall Officials: Tarık EMre Sener, Assoc. Prof., Principal Investigator — Marmara University, School of Medicine, Department of Urology
Locations (1):
- Marmara University, School of Medicine, Department of Urology, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Upon request, study data can be shared without sharing participant identifying personal data.

REFERENCES:
- [Background] Tang J, Yang JC, Zhang Y, Liu X, Zhang L, Wang Z, Li J, Luo Y, Xu J, Shi H. Does benign prostatic hyperplasia originate from the peripheral zone of the prostate? A preliminary study. BJU Int. 2007 Nov;100(5):1091-6. doi: 10.1111/j.1464-410X.2007.07081.x. PMID 17922787
- [Background] Chughtai B, Forde JC, Thomas DD, Laor L, Hossack T, Woo HH, Te AE, Kaplan SA. Benign prostatic hyperplasia. Nat Rev Dis Primers. 2016 May 5;2:16031. doi: 10.1038/nrdp.2016.31. PMID 27147135
- [Background] Dahm P, Brasure M, MacDonald R, Olson CM, Nelson VA, Fink HA, Rwabasonga B, Risk MC, Wilt TJ. Comparative Effectiveness of Newer Medications for Lower Urinary Tract Symptoms Attributed to Benign Prostatic Hyperplasia: A Systematic Review and Meta-analysis. Eur Urol. 2017 Apr;71(4):570-581. doi: 10.1016/j.eururo.2016.09.032. Epub 2016 Oct 4. PMID 27717522
- [Background] Plochocki A, King B. Medical Treatment of Benign Prostatic Hyperplasia. Urol Clin North Am. 2022 May;49(2):231-238. doi: 10.1016/j.ucl.2021.12.003. Epub 2022 Mar 22. PMID 35428429
- [Background] Cornu JN, Zantek P, Burtt G, Martin C, Martin A, Springate C, Chughtai B. Minimally Invasive Treatments for Benign Prostatic Obstruction: A Systematic Review and Network Meta-analysis. Eur Urol. 2023 Jun;83(6):534-547. doi: 10.1016/j.eururo.2023.02.028. Epub 2023 Mar 22. PMID 36964042
- [Background] Franco JVA, Jung JH, Imamura M, Borofsky M, Omar MI, Escobar Liquitay CM, Young S, Golzarian J, Veroniki AA, Garegnani L, Dahm P. Minimally invasive treatments for benign prostatic hyperplasia: a Cochrane network meta-analysis. BJU Int. 2022 Aug;130(2):142-156. doi: 10.1111/bju.15653. Epub 2021 Dec 6. PMID 34820997
- [Background] He W, Ding T, Niu Z, Hao C, Li C, Xu Z, Jing Y, Qin W. Reoperation after surgical treatment for benign prostatic hyperplasia: a systematic review. Front Endocrinol (Lausanne). 2023 Nov 9;14:1287212. doi: 10.3389/fendo.2023.1287212. eCollection 2023. PMID 38027158
- [Background] Magistro G, Schott M, Keller P, Tamalunas A, Atzler M, Stief CG, Westhofen T. Enucleation vs. Resection: A Matched-pair Analysis of TURP, HoLEP and Bipolar TUEP in Medium-sized Prostates. Urology. 2021 Aug;154:221-226. doi: 10.1016/j.urology.2021.04.004. Epub 2021 Apr 21. PMID 33891930
- [Background] Mavuduru RM, Mandal AK, Singh SK, Acharya N, Agarwal M, Garg S, Kumar S. Comparison of HoLEP and TURP in terms of efficacy in the early postoperative period and perioperative morbidity. Urol Int. 2009;82(2):130-5. doi: 10.1159/000200786. Epub 2009 Mar 19. PMID 19321996
- [Background] Chavali JSS, Rivera ME, Lingeman JE. HoLEP Learning Curve-Resident Perspective: Survey of Senior Residents from High-Volume Tertiary Center. J Endourol. 2024 Sep;38(9):977-981. doi: 10.1089/end.2024.0054. Epub 2024 Jul 4. PMID 38904168
- [Background] Wenk MJ, Hartung FO, Egen L, Netsch C, Kosiba M, Grune B, Herrmann J. The long-term learning curve of holmium laser enucleation of the prostate (HoLEP) in the en-bloc technique: a single surgeon series of 500 consecutive cases. World J Urol. 2024 Jul 24;42(1):436. doi: 10.1007/s00345-024-05097-9. PMID 39046537
- [Background] Martinez-Salas AJ, Garcia-Rivera OU, Reyna-Blanco I, Jimenez-Garcia AD, Rosas-Hernandez H. Adequate Mentorship Program for Holmium Laser Enucleation of the Prostate (HoLEP) Leads to Satisfactory Short-Term Outcomes in the Early Learning Curve of Young Urologists: First-Year Outcomes of a Newly Established Mentorship Training in Mexico. Cureus. 2023 Jul 12;15(7):e41756. doi: 10.7759/cureus.41756. eCollection 2023 Jul. PMID 37575804
- [Background] Baron M, Nouhaud FX, Delcourt C, Grise P, Pfister C, Cornu JN, Sibert L. [HoLEP learning curve: Toward a standardised formation and a team strategy]. Prog Urol. 2016 Sep;26(9):492-9. doi: 10.1016/j.purol.2016.08.002. Epub 2016 Sep 7. French. PMID 27614386